CLINICAL TRIAL: NCT06289166
Title: A Multi-center, Open-label, Phase Ⅱb Trial to Evaluate the Safety and Efficacy of STSP-0601 for Injection in Patients with Hemophilia with Inhibitor
Brief Title: Safety and Efficacy of STSP-0601 in Adult Patients with Hemophilia a or B with Inhibitor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STSP-0601-04
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Consecutive doses of STSP-0601 (Experimental)
  Interventions: Drug: STSP-0601 for Injection

INTERVENTIONS:
Drug: STSP-0601 for Injection — A Multiple-dose Design to Evaluate the Safety, Tolerability and Efficacy of STSP-0601 for Injection in hemophilia A or B patients with inhibitor.

SUMMARY:
This study will assess the safety and efficacy of multiple-dose of STSP-0601 for the treatment of bleeding episodes in hemophilia A or B patients with inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. 18 ≤age≤70 years of age,male.
2. Hemophilia A or B patients. (No less than 3 patients with hemophilia B)
3. Peak historical inhibitor titer ≥ 5 BU and apositive inhibitor test when enrolled.
4. Establish proper venous access.
5. There were at least 3 bleeding events that requiring treatment occurred in the past 6 months before screening (Only applicable to the on-demand treatment stage).
6. Agree to use adequate contraception to avoid pregnancy. Agree not to donate sperm or eggs.
7. Provide signed informed consent.

Exclusion Criteria:

1. Have any coagulation disorder other than hemophilia.
2. Plan to receive prophylactic treatment of coagulation factor during the trail.
3. Patients plan to receive Emicizumab during the trial.
4. Patients received anticoagulant or antifibrinolytic therapy 7 days before enrollment or plan to receive these drugs during the trial.Patients received anticoagulation therapy (such as coagulation factor replacement therapy, prothrombin complex, plasma, etc.) 7 days before enrollment.
5. Have a history of arterial and/or venous thrombotic events.
6. Platelet <100×109/L.
7. Hemoglobin<90g/L.
8. Severe liver or kidney disease.
9. Severe bleeding event occurred within 4 weeks before enrollment.
10. Accepted major operation or blood transfusion within 4 weeks before enrollment.
11. Have a known allergy to STSP-0601.
12. Pregnant, lactating, or blood pregnancy test positive female subjects
13. Participate in other clinical research within 4 weeks before enrollment(except for participating in prothrombin complex, FVII, FVIIa, FVIII, FIX trails).
14. Within 1 day prior to enrollment, FVII, FVIIa, tranexamic acid, and aminocaproic acid were used. Within 3 days prior to enrollment, prothrombin complex, FVIII, and FIX were used. Within 4 weeks prior to enrollment, treatment with amisulumab was received.
15. Patients not suitable for the trail according to the judgment of the investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Proportion of successfully treated bleeding episodes | 12 hours after first administration of study drug

SECONDARY OUTCOMES:
Proportion of successfully treated first bleeding episodes | 12 hours after first administration of study drug
Proportion of successfully treated bleeding episodes | 8 hours after first administration of study drug
Excellent + good rate of treated bleeding episodes | 12 hours after first administration of study drug
  Excellent: Pain and Symptoms of bleed (e.g., swelling, tenderness, and decreased range of motion in the case of musculoskeletal haemorrhage) had fully eased. No additional infusion of study drug was required.
  Good: Symptoms of bleed (e.g., swelling, tenderness, and decreased range of motion in the case of musculoskeletal haemorrhage) had largely eased , but had not completely disappeared. No additional infusion of study drug was required.
Excellent + good rate of treated bleeding episodes | 8 hours after first administration of study drug
  Excellent: Pain and Symptoms of bleed (e.g., swelling, tenderness, and decreased range of motion in the case of musculoskeletal haemorrhage) had fully eased. No additional infusion of study drug was required.
  Good: Symptoms of bleed (e.g., swelling, tenderness, and decreased range of motion in the case of musculoskeletal haemorrhage) had largely eased , but had not completely disappeared. No additional infusion of study drug was required.
Number of doses required for effective hemostasis | 12 hours after first administration of study drug
Proportion of bleeding episodes received salvage treatment | 24 hours after first administration of study drug
Time to complete/significant remission from first dose | 72 hours after last administration of study drug
Time to complete/significant remission from haematogenesis | 72 hours after last administration of study drug
Proportion of successfully treated Target joint bleeding episodes | 12 hours after first administration of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, Ph.D, Principal Investigator — Hospital of Hematology, Chinese Academy of Medical Sciences
Locations (20):
- China (20):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Affiliated Union Medical College Hospital, Fuzhou, Fujian
  - Lanzhou University First Hospital, Lanzhou, Gansu
  - Southern Medical University Southern Hospital, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Guizhou Medical University Affiliated Hospital, Guiyang, Guizhou
  - Harbin First Hospital Hematology Tumor Research Center, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing University School of Medicine Affiliated Gulou Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The first hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital Affiliated to China Medical University, Shenyang, Liaoning
  - Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Xi'an Central Hospital, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Hospital of Hematology, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu W, Zhou H, Huang R, Du X, Wang P, Zhou Z, Zheng C, Lou S, Ma J, Song Y, Dai X, Wang X, Yang R, Zhang L. A specific FX activator for bleeding treatment in hemophilia with inhibitors: multicenter, open-label, phase I/II trials. Blood Adv. 2026 Feb 4:bloodadvances.2025019486. doi: 10.1182/bloodadvances.2025019486. Online ahead of print. PMID 41637644